CLINICAL TRIAL: NCT05676697
Title: Safety and Efficacy Study of PI3K Delta Inhibitor in Relapsed / Refractory Autoimmune Hemolytic Anemia Patients After Receiving Two or More Lines of Therapy
Brief Title: PI3K Delta Inhibitor in Relapsed / Refractory Autoimmune Hemolytic Anemia Patients After Receiving Two or More Lines of Therapy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Did not meet the anticipated outcome.
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: YL-Pharma (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2022067
Record Dates: First submitted 2022-12-07; First posted 2023-01-09 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2024-02

CONDITIONS: Autoimmune Hemolytic Anemia; Failure of Two Rounds of Treatment
MeSH Terms: conditions — Anemia, Hemolytic, Autoimmune

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PI3K Delta Inhibitor (Experimental)
  Interventions: Drug: Linperlisib

INTERVENTIONS:
Drug: Linperlisib — The phosphatidylinositol 3-kinase delta (PI3Kδ) signaling pathway plays a critical role in the activation, proliferation, and tissue homing of self-reactive B cells that contribute to autoimmune diseases. B cells play an essential role in immune system function and dysfunction (e.g., autoimmunity) by producing antibodies and by acting as antigen-presenting cells (APCs) for T cells. Signaling via PI3K controls many essential B cell functions and is therefore a promising target for preventing aberrant B cell activation.

SUMMARY:
This is a prospective, multicenter, single-arm, pilot study. The aim of this study is to evaluate the efficacy and safety of Linperlisib, the PI3K delta inhibitor for autoimmune hemolytic anemia patients who failed the second line therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age ≥ 18 years
* Diagnosis of primary warm antibody hemolytic anemia (AIHA).
* Hemoglobin < 100g/L
* Refractory to or relapsed after at least 2 prior treatment line.
* ECOG performance status ≤ 2
* Willing and able to comply with the requirements for this study and written informed consent.

Exclusion Criteria:

* Neutrophils counts < 0.5×10^9/L or platelet counts < 50 x 10^9/L
* Diagnosis of any of the following diseases: Cold agglutinin disease, cold agglutinin syndrome, mixed AIHA, paroxysmal cold hemoglobinuria (PCH).
* Diagnosis of the active stage of the connective tissue or systemic autoimmune rheumatic diseases (SARDs)
* History of lymphoproliferative neoplasms
* Had other inherited or acquired hemolytic diseases.
* Secondary AIHA caused by drugs or infection
* Previously received organ or stem cell transplantation.
* Had malignant tumor within 5 years before enrollment, exclusive of cured basal or squamous cell skin cancer, superficial bladder cancer, prostate intraepithelial tumor, cervical carcinoma in situ or other indolent tumors
* Patients with HBV, HCV, HIV or other infections that require treatment.
* Abnormal liver function: two consecutive examinations with an interval of ≥1 week suggest that ALT and AST are 2.5 times higher than the upper limit of normal values
* Renal impairment: creatinine clearance <60ml/min
* Any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study, including clinically significant cardiac diseases, refractory hypertension, metabolic disorders and other diseases that seriously affect the function of the gastrointestinal tract.
* Had a history of any psychiatric diseases, cerebrovascular disease or cognitive sequelae of head injury.
* Received rituximab in 6 weeks before enrollment.
* Received attenuated vaccine 4 in weeks before enrollment
* Participation in another clinical trial within 4 weeks before the start of this trial
* Have an allergy to Linperlisib or any other part of this medicine.
* Previously treated with other PI3Kδ inhibitor.
* Pregnant or breast-feeding patients
* Patients considered to be ineligible for the study by the investigator for reasons other than the above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-01-13 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-02-06 (Actual)

PRIMARY OUTCOMES:
Overall response rate | 6-12 weeks
  Percentage of patients with hematological response. Hematological response is evaluated by hemoglobin and other hemolysis-related laboratory indicators.

SECONDARY OUTCOMES:
Incidence of the adverse event | 12 weeks
  Use Common Terminology Criteria for Adverse Events (CTCAE) Version 5 to assess the adverse event.
Complete response rate | 6-12 weeks
  Percentage of patients with hematological complete response. Hematological response is evaluated by hemoglobin and other hemolysis-related laboratory indicators.
Complete response with incomplete hemolysis recovery, CRi | 6-12 weeks
  Percentage of patients with CRi which is evaluated by hemoglobin and other hemolysis-related laboratory indicators.
Mean change from baseline in hemoglobin (Hgb) levels | 6-12 weeks
Time to achieve partial response (PR) | 6-12 weeks
  Duration time was calculated from enrollment to PR. PR is assessed by hemoglobin and blood transfusion.
Time to achieve complete response (CR) | 6-12 weeks
  Duration time was calculated from enrollment to CR.
Change of the health-related quality of life | Baseline and 12 weeks
  Medical Outcomes Study Questionnaire Short Form 36 Health Survey (SF-36) is used to assess the health-related quality of life of patients. The SF-36 has eight scaled scores; the scores are weighted sums of the questions in each section. Scores range from 0 - 100. Lower scores = more disability, higher scores = less disability

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Zhoukou Central Hospital, Zhoukou, Henan
  - Regenerative Medicine Center, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No